CLINICAL TRIAL: NCT02776631
Title: Pinloc Versus Hansson Pins in the Treatment of Femoral Neck Fractures: A Prospective Randomized Study of 500 Patients
Brief Title: Pinloc Versus Hansson Pins in the Treatment of Femoral Neck Fractures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Torsten Johansson (Other)
Collaborators: Sahlgrenska University Hospital (Other); Department of Orthopedics, Motala (Unknown); Department of Orthopedics, Norrköping (Unknown); Department of Orthopedics, Nykoeping (Unknown); Department of Orthopedics, Eskilstuna (Unknown); Department of Orthopedics, Falun (Unknown); Department of Orthopedics, Uppsala University Hospital (Unknown); Department of Orthopedics, Helsingborg (Unknown)
Responsible Party: Sponsor-Investigator, Torsten Johansson, MD (Orthopedic surgeon), Associate professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pinloc study
Record Dates: First submitted 2016-01-20; First posted 2016-05-18 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pinloc (Experimental): Plate and 3 interlocked pins. A new device for fixation of femoral neck fractures.
  Interventions: Device: Pinloc
- LIH (Hansson pins) (Active Comparator): 2 pins. An established method for fixation of femoral neck fractures.
  Interventions: Device: Hansson Pins (LIH)

INTERVENTIONS:
Device: Pinloc — Internal fixation device
  Arms: Pinloc
Device: Hansson Pins (LIH) — Internal fixation device
  Arms: LIH (Hansson pins)

SUMMARY:
A prospective randomized study comparing a new implant with three interlocked pins for internal fixation of femoral neck fractures (Hansson Pinloc System, Swemac Linköping, Sweden) versus 2 parallel pins with hooks (Hansson Pins, Swemac Linköping, Sweden).

DETAILED DESCRIPTION:
Patients, who are to be treated with internal fixation due to a femoral neck fracture, will be randomized by the surgeon to Pinloc or Hansson Pins using an on-line randomization system.

The patients will be followed up at open visits at 3 months and 1 year. At two years the patients will be contacted by phone and medical records studied in order to detect any fracture complications.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fractures where the preferred treatment is internal fixation.

Exclusion Criteria:

* Unwilling to participate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Failure of fracture treatment | Within 2 years postoperatively
  Failure is defined as non-union or avascular necrosis.

SECONDARY OUTCOMES:
Timed-up and go test | At 3 months and 1 year postoperatively
  Stand up, walk 3 meters, turn around and sit down
WOMAC (An established hip score) | At 3 months and 1 year postoperatively
  An established hip score
Quality of life (EQ-5D) | At 3 months and 1 year postoperatively
  EQ-5D
Pain (Visual analogue scale) | At 3 months and 1 year postoperatively
  Visual analogue scale (VAS): At rest and during activity

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Johansson, MD,Ass prof, Principal Investigator — Division of Orthopaedics, Department of Clinical and Experimental Medicine, Faculty of Health Sciences, Linköping University, Sweden.; Torsten Johansson, MD,Ass prof, Study Director — Division of Orthopaedics, Department of Clinical and Experimental Medicine, Faculty of Health Sciences, Linköping University, Sweden.
Locations (8):
- Sweden (8):
  - Department of Orthopedics, Eskilstuna
  - Department of Orthopedics, Falun
  - Department of Orthopaedics, Gothenburg
  - Department of Orthopedics, Helsingborg
  - Department of Orthopedics, Aleris, Motala
  - Department of Orthopedics, Norrköping
  - Department of Orthopedics, Nyköping
  - Department of Orthopedics, Uppsala

IPD SHARING:
Plan to Share IPD: Yes